CLINICAL TRIAL: NCT07333495
Title: A Mixed Cohort, Multicentre Exploratory Study of Non-invasive Quantitative Assessment of Renal Graft Function With Non-contrast Functional Magnetic Resonance Imaging
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Zhen Li, Professor, Tongji Hospital
Other Study IDs: TJ-IRB202512022; TJ-IRB202512022 (Other: Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology Department of Radiology)
Record Dates: First submitted 2025-12-12; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Kidney Transplant; Renal Allograft Recipients; Renal Allograft
Keywords: renal allograft; MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paired Donor-Recipient Cohort: Kidney transplant recipients enrolled along with their corresponding donor (living or deceased). The donor undergoes a pre-transplant MRI to establish an individualized functional baseline for the graft. This cohort aims to achieve ultra-sensitive detection of post-transplant functional changes by comparing against the kidney's own baseline.
- Independent Recipient Cohort: Kidney transplant recipients for whom donor baseline data is unavailable (primarily recipients of deceased donor kidneys). This cohort is used to validate the standalone capability of the non-contrast MRI protocol for monitoring graft function dynamics over time, addressing the common clinical scenario where donor information is absent.

SUMMARY:
This clinical study aims to investigate a new, non-invasive method for monitoring kidney function after transplantation. Currently, assessing the health of a transplanted kidney often relies on blood tests or invasive biopsies, which may not detect subtle early changes or account for each kidney's unique starting point.

This research will use advanced, non-contrast Magnetic Resonance Imaging (MRI) scans to measure various aspects of kidney health, such as blood flow and oxygen levels. The study includes two main groups of participants: 1) kidney transplant donors and their matched recipients, and 2) transplant recipients whose donors are unavailable for study (e.g., deceased donors).

For donor-recipient pairs, the goal is to create a personalized "baseline" for each transplanted kidney by scanning the donor before donation. This allows doctors to compare the kidney's function after transplant to its own unique starting point, potentially detecting problems much earlier. For recipients without donor data, the study will evaluate how well the MRI scans can track changes in kidney function over time on their own.

Additionally, the study will analyze body composition (like fat and muscle distribution) and metabolic health to understand their relationship with transplant kidney function. We plan to enroll approximately 1000 participants across multiple hospitals. The ultimate goal is to develop a more accurate, individualized, and non-invasive tool for the early detection of transplant kidney problems, helping to improve long-term outcomes and quality of life for transplant patients.

DETAILED DESCRIPTION:
This is a prospective, multicenter, hybrid cohort study designed to validate a non-contrast functional MRI protocol for the non-invasive, quantitative assessment of graft function in kidney transplant recipients.

Primary Objectives:

To establish an individualized functional baseline for transplanted kidneys through donor-recipient paired studies, moving beyond population-based reference values to enable a "self-comparison" paradigm for enhanced sensitivity in detecting early graft dysfunction.

To validate the standalone capability of non-contrast functional MRI for sensitively monitoring dynamic changes in graft function in a large, independent cohort of recipients without donor baseline data (e.g., from deceased donors).

To integrate MRI parameters with body composition analysis and metabolic profiles to build a comprehensive, non-invasive assessment model for early diagnosis, treatment evaluation, and prognosis prediction of graft function.

Study Cohorts:

Paired Study Cohort: Live or deceased kidney transplant donors who can undergo pre-transplant baseline MRI and their corresponding recipients.

Independent Recipient Cohort: Kidney transplant recipients for whom donor baseline data is unavailable (primarily from deceased donors).

Key Assessments:

MRI Protocol: Includes multiple non-contrast functional sequences (e.g., DWI, ASL, BOLD, MT) to quantitatively evaluate renal perfusion, oxygenation, diffusion, and microstructure.

Clinical & Laboratory Data: Collection of serial serum creatinine, eGFR, uric acid, proteinuria, and other relevant biomarkers.

Body Composition Analysis: MRI-based quantification of visceral, subcutaneous, perirenal, sinus renalis fat, and muscle mass.

Histopathology: When available, biopsy results (e.g., rejection classification, fibrosis scores) will be collected as a reference standard.

Study Procedures: Eligible participants will undergo non-contrast MRI scans at scheduled follow-up visits. Clinical data, laboratory results, and body composition metrics will be collected concurrently. For the paired cohort, donor baseline MRI (pre-transplant) serves as the individual reference. All data will be anonymized and analyzed to correlate MRI parameters with clinical, laboratory, and histopathological outcomes.

Sample Size: The planned sample size is 1000 participants. This calculation is based on the inclusion of approximately 80 potential predictor variables (from MRI, clinical, and metabolic data) for multivariate analysis, requiring a sample size at least 10 times the number of variables, with an additional allowance for a 20% drop-out rate.

Potential Impact: This study seeks to provide a novel, practical, and individualized solution for the precise monitoring of transplant kidney function, addressing a critical unmet need in clinical management, particularly for recipients of deceased donor organs.

ELIGIBILITY:
Inclusion Criteria:

Adult participants (age ≥ 18 years).

For the Paired Donor-Recipient Cohort:

Donor: Scheduled for living kidney donation, OR is a deceased organ donor who can undergo a pre-transplant MRI.

Recipient: Recipient of a kidney transplant or simultaneous pancreas-kidney transplant from the paired donor.

For the Independent Recipient Cohort:

Recipient: Recipient of a kidney transplant from a deceased donor for whom donor baseline data is unavailable.

Able to provide informed consent.

Exclusion Criteria:

Any contraindication to MRI (e.g., cardiac pacemaker, non-MRI compatible metallic implants, neurostimulators, severe claustrophobia).

Inability to tolerate the breath-holding required for MRI acquisition.

Pregnancy.

Any clinical condition that, in the investigator's judgment, would severely compromise study participation or data integrity (e.g., uncontrolled severe infection, active major psychiatric illness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll adult (age ≥18 years) kidney transplant recipients and their corresponding donors from multiple participating transplant centers.
  This hybrid cohort comprises two distinct sub-populations:
  Paired Donor-Recipient Cohort: Includes both the transplant recipient and the living or deceased donor from whom the kidney originated.
  Independent Recipient Cohort: Includes transplant recipients (primarily from deceased donors) for whom paired donor baseline data is not available.
  All enrolled participants will undergo a standardized, non-contrast functional MRI assessment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Functional MRI for pathology in Kidney Transplant Recipients (Including T-Cell Mediated and Antibody-Mediated Rejection) | From the time of transplantation hospitalization until the end of the study follow-up period (up to 5 years). Assessments will be performed at each time point where a transplant kidney biopsy is deemed necessary by the clinician
  At the time of each clinically indicated biopsy, the required data (e.g., for functional MRI) will be collected. The results will be compared against the reference standard of histopathological diagnosis from the concurrent transplant kidney biopsy, graded according to the updated Banff classification criteria. The primary analysis will be the diagnostic sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV), each presented with a 95% confidence interval. Secondary analysis will include the correlation between the functional MRI findings and the severity grade of Banff lesions.

SECONDARY OUTCOMES:
Correlation between Baseline Functional MRI Parameters and Long-Term Decline in Renal Allograft Function | From the first functional MRI assessment post-transplant, with subsequent assessments of renal function at Years 1, 2, 3, 4, and 5.
  Functional MRI parameters (e.g., derived from sequences such as BOLD, DWI, or DTI) obtained at the baseline post-transplant assessment will be analyzed. Their association with the longitudinal change in graft function will be evaluated. Graft function will be primarily assessed by the estimated glomerular filtration rate (eGFR). The rate of renal function decline will be quantified (e.g., as the annualized slope of eGFR change over the 5-year follow-up period). The strength of the correlation/association will be calculated using appropriate statistical methods (e.g., Pearson's or Spearman's correlation coefficient, or linear mixed-effects models), with a significance level set at p < 0.05.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Sinopharm Dongfeng General Hospital, Dongfeng Motor Corporation and Hubei University of Medicine., Shiyan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Shanxi Bethune Hospital, Shanxi Academy of Medical Sciences, Shanxi Medical University, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No
protect patient privacy